CLINICAL TRIAL: NCT01428349
Title: Matching Cognitive Remediation to Cognitive Deficits in Substance-Abusing Inmates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SE-2011-0103
Record Dates: First submitted 2011-08-17; First posted 2011-09-05 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2011-11

CONDITIONS: Psychopathy; Personality Disorders
Keywords: Incarcerated offenders; emotionally reactive; emotionally stable; psychopathy
MeSH Terms: conditions — Antisocial Personality Disorder; Personality Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention to Context (Experimental)
  Interventions: Other: Cognitive Remediation
- Affective Cognitive Control (Experimental)
  Interventions: Other: Cognitive Remediation

INTERVENTIONS:
Other: Cognitive Remediation — Computer training on 3 tasks that targets the attention to context deficits associated with psychopathic offenders. Participants complete 6 training sessions, that include the tasks, feedback and real-world translational examples.
  Arms: Attention to Context
Other: Cognitive Remediation — Computer training on 3 tasks that targets the affective cognitive control deficits associated with externalizing offenders. Participants complete 6 training sessions, that include the tasks, feedback and real-world translational examples.
  Arms: Affective Cognitive Control

SUMMARY:
This is a 2 -year NIDA funded grant (Co-PIs: Joseph P. Newman, John Curtin, and Carl Lejuez) that examines whether recent progress in characterizing the cognitive deficits associated with psychopathic and externalizing offenders may be used to develop better therapeutic interventions to treat their substance abuse and other self-control problems. Inmates with externalizing or psychopathy will receive one of two computer-based interventions to remediate the core cognitive skills that have been linked to self-regulation deficits in the two groups. One intervention (ACC) targets the affective cognitive control deficits associated with externalizing offenders whereas the other intervention (ATC) targets the attention to context deficits associated with psychopathic offenders. The specific components of the project include: selection and randomization of inmates; pre- and post-treatment behavioral and brain-related (ERP and Startle) measures to evaluate the impact and specificity of the ACC and ATC treatments; and 6 sessions of behavioral (e.g. computerized) and verbal training in ACC or ATC.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* ages 18-45 years,
* elevated scores of psychopathy or externalizing measures

Exclusion Criteria:

* currently taking psychotropic medication,
* below a 4th grade reading level,
* history or current learning disability,
* history of head trauma with lasting effects,
* current diagnosis of PTSD,
* Bipolar, or
* psychosis

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Psychophysiological change from pre-treatment to post-treatment | 6 weeks after pre-testing
  We will measure electrophysiology (EEG), startle responses (EMG measured in microvolts), and behavioral responses on six tasks that measure such processes as affective regulation, distress tolerance, cognitive control, selective attention, and attending to context.

SECONDARY OUTCOMES:
Frequency of Conduct Reports | within 3 months of participation
  Assess change in the frequency of institution conduct reports post-treatment. We will compare frequency of these reports pre-treatment and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Newman, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Fox Lake Correctional Institution, Fox Lake, Wisconsin
  - Oshkosh Correctional Institution, Oshkosh, Wisconsin

REFERENCES:
- [Result] Baskin-Sommers AR, Curtin JJ, Newman JP. Altering the Cognitive-Affective Dysfunctions of Psychopathic and Externalizing Offender Subtypes with Cognitive Remediation. Clin Psychol Sci. 2015 Jan 1;3(1):45-57. doi: 10.1177/2167702614560744. PMID 25977843